CLINICAL TRIAL: NCT03858608
Title: A Pragmatic, Randomised, Controlled, Trial of the Effect of the Counterweight Plus Weight Management Programme in Uncontrolled Asthma Associated With Elevated Body Mass Index
Brief Title: Weight Loss for Uncontrolled Asthma Associated With Elevated BMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GN18RM508
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Asthma; Obesity
Keywords: Weight loss; Counterweight Plus
MeSH Terms: conditions — Asthma; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Unblinded, pragmatic, pilot, randomised, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counterweight Plus (Experimental): Total Diet Replacement phase (0-12 weeks) 825-853kcal/day low energy liquid diet (LELD) for 12 weeks Food Reintroduction phase (13-18 weeks) Wk 13: 400kcal/d LELD + 1 low-fat meal/day (c. 360-400 kcal) + 2 servings of fruit, 200mls skimmed milk and free vegetables. Total intake: 1000kcal/day Wk 15: 200kcal/d LELD + 2 low-fat meals/day (c. 720-800 kcal) + 2 servings of fruit, 200mls skimmed milk and free vegetables. Total intake: 1200kcal/day.
  Wk 17: 3 low-fat meals per day (c.1080-1200 kcal) + 2 servings of fruit, 200mls skimmed milk and free vegetables. Total intake: 1400kcal/day.
  Weight maintenance phase (wks 19-52) Low-fat healthy eating weight loss maintenance intervention [target below 30% energy from fat, with flexibility to optimise individual compliance, to a maximum of 35%]
  Interventions: Dietary Supplement: Counterweight Plus
- Usual asthma care (Active Comparator): Usual asthma management
  Interventions: Other: Usual asthma care

INTERVENTIONS:
Dietary Supplement: Counterweight Plus — Total diet replacement followed by food reintroduction and weight maintenance.
  Arms: Counterweight Plus
Other: Usual asthma care — Usual asthma management
  Arms: Usual asthma care

SUMMARY:
Weight loss for uncontrolled asthma associated with elevated BMI. Asthma is a common condition with different types recognised that have variable responses to current treatments. It is often poorly controlled and there is a need to discover new treatments. Obesity is common in asthma and is associated with increase in symptoms, poorer asthma control and quality of life, and increased healthcare utilisation and treatment burden. The Counterweight Plus programme is a safe, evidence-based non-surgical intervention that is associated with sustained weight losses of up to 15% in obese individuals but its effects in asthma have not been tested. Our study aims to evaluate the impact of this intervention in individuals with difficult asthma associated with obesity.

The Counterweight Plus programme includes a total diet replacement (TDR) phase (12 weeks) followed by structured food reintroduction (6 weeks) and long term weight loss maintenance (34 weeks) and will be provided by Dieticians trained in the delivery of this intervention. Participants will attend fortnightly clinic reviews with Dieticians during the first 18 weeks and then monthly clinic reviews during the weight loss maintenance period.

Participants will be randomised to Counterweight Plus programme or usual care (control) and followed for 1 year with study visits at baseline, 4 months and 1 year. During study visits participants will be invited to complete questionnaires, provide a blood sample, perform breathing tests and a walking test, and wear an activity monitor for one week.

If the Counterweight Plus programme is proven to be of benefit in this patient group, this may lead to service development so that this intervention may be made available to similar patients in the future within the clinical setting.

DETAILED DESCRIPTION:
This study will be a unblinded, pragmatic, pilot, randomised, controlled trial of the Counterweight Plus programme versus usual care in individuals with difficult asthma associated with obesity. Eligible individuals will be identified through Difficult Asthma Clinics or ward admissions. Those wishing to participate will receive an information sheet and be invited to provide written informed consent prior to commencing the study.

Baseline Visit

Measurements taken at the baseline visit will include:

Demographics - age, gender, smoking history (current, ex, none, years since stopped, pack years), age at asthma diagnosis, duration of asthma, atopy, co-morbidities (allergic/perennial rhinitis, nasal polyps, nasal surgery, eczema, gastro-oesophageal reflux disease, diabetes, hypertension, cardiac disease, osteopenia/osteoporosis etc), medications (inhaled/nebulised short acting beta2-agonists (SABA), inhaled and oral corticosteroids etc), healthcare usage (oral corticosteroid (OCS) boosts, unscheduled General Practitioner (GP) or Accident + Emergency (A+E) attendances, hospital and Intensive Care Unit (ICU) admissions in preceding year), weight, height and BMI.

Questionnaires - Medical Research Council (MRC) dyspnoea scale, Asthma Control Questionnaire (ACQ6), Asthma Quality of Life Questionnaire (AQLQ), and Hospital Anxiety and Depression Scale (HAD).

Venepuncture - full blood count, urea and electrolytes, liver function tests, magnesium, bone profile, insulin, glucose, HbA1c, lipids, C-reactive Protein (CRP), Interleukin-6 (IL-6), leptin and adiponectin Lung Function/inflammometry - peak expiratory flow (PEF) (best of 3), Spirometry (pre- and post-bronchodilator), Fraction of exhaled nitric oxide (FENO) Exercise tolerance - 6 minute walk test (practice test and repeat test)[29], Modified Borg Dyspnoea Scale, pulse oximetry.

Physical Activity - actigraphy. Participants will be given the Actigraph device and asked to wear it continuously for 7 days on their non-dominant wrist, then hand it back.

Participants will be provided with a Personalized Asthma Management Plan, and Symptoms Diary that includes SABA use and other healthcare usage (oral corticosteroid (OCS) boosts, unscheduled GP or A+E attendances, hospital and ICU admissions); inhaler technique will be corrected if necessary.

Participants will be randomized 1:1 to Group A and Group B. Group A will enter the Counterweight Plus programme and Group B will enter the usual care arm.

Participants will return for Visit 2 at 16 weeks and Visit 3 at 52 weeks.

Measurements taken at Visits 2 and 3 will include:

Demographics - medications (inhaled/nebulised short acting beta2-agonists (SABA), inhaled and oral corticosteroids etc), healthcare usage (oral corticosteroid (OCS) boosts, unscheduled GP or A+E attendances, hospital and ICU admissions since last visit), weight, height, and BMI.

Questionnaires - MRC dyspnoea scale, Asthma Control Questionnaire (ACQ6), Asthma Quality of Life Questionnaire (AQLQ), and Hospital Anxiety and Depression Scale (HAD).

Venepuncture - full blood count, urea and electrolytes, liver function tests, magnesium, bone profile, insulin, glucose, HbA1c, lipids, CRP, IL-6, leptin and adiponectin Lung Function/inflammometry - PEF (best of 3), Spirometry (pre- and post-bronchodilator), Fraction of exhaled nitric oxide (FENO) Exercise tolerance - 6 minute walk test, Modified Borg Dyspnoea Scale, pulse oximetry.

Physical Activity - actigraphy Visits will be postponed by 4 weeks in the event of exacerbation or respiratory infection. Throughout the study period changes to asthma medications will be allowed as clinically indicated.

Rescue Package for weight regain or re-emergence of diabetes Some patients find weight maintenance difficult, some relapse temporarily and gain weight rapidly. Others may tend to let things slip more gradually. Pilot studies showed the value of a sympathetic, but firm approach to relapse/regain management. If weight regains occurs in TDR randomised participants, or if diabetes is found to have returned (HbA1c risen above 6.5%) at any time during the 18 month weight loss maintenance stage, 'rescue plans' for weight gain prevention will be offered.

1. Weight regain of >2kg: offer the use of TDR to replace one main-meal per day for 4 weeks, and offer orlistat 120 mg tid, with each meal.
2. Weight gain of >4kg, or to <15kg below starting weight or if diabetes recurs: offer 4 weeks TDR with fortnightly weekly practice nurse/dietitian review and then a 2-4 week food re-introduction (adding 1 meal/week as before). Lowfat dietary advice and physical activity will be reinforced for weight maintenance and orlistat treatment will be offered.

This package can be repeated as required in each year of the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed asthma as per Global Initiative for Asthma (GINA) guidelines 2015 with characteristic symptoms and at least one of the following:

   • Reversible airflow limitation - 12% and 200ml increase in forced expiratory volume (FEV1) in the preceding 5 years either: i. After inhaled/nebulised bronchodilator or 4+ weeks of anti-inflammatory treatment ii. Between visits

   • Positive bronchial challenge in the preceding 5 years: i. Provocation concentration (PC20) methacholine or histamine <8mg/ml ii. Provocative dose (PD15) mannitol <635mg
2. Difficult asthma defined as per Scottish Intercollegiate Guidelines Network (SIGN)/British Thoracic Society (BTS) guideline 2014 as persistent symptoms and/or frequent asthma attacks despite treatment at step 4 or step 5 with either:

   * ACQ6 >1.5
   * ≥2 systemic corticosteroid boosts in previous year
   * ≥1 hospitalization in previous year
3. BMI ≥ 30 kg/m2

Exclusion Criteria:

1. ICU admission +/- mechanical ventilation in the previous 6 months for asthma exacerbation
2. Respiratory tract infection requiring antibiotics or asthma exacerbation requiring corticosteroid boost in preceding 4 weeks
3. Significant respiratory or other co-morbidity likely to influence the conduct of the study
4. Pregnancy and breast feeding
5. Severe and/or unstable cardiac disease
6. Recent (within the preceding 6 months) commencement of antifungal, biologic (omalizumab, lebrikizumab, mepolizumab) or "Airsonett" device; eligible if on treatment for > 6months or discontinued
7. Current insulin use
8. Current treatment with anti-obesity drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Asthma Control overall change | Baseline to week 16
  Change in score of ACQ6 (Asthma Control Questionnaire 6) in intervention group versus usual care group. Score range 0 - 36 with higher scores representing a worse outcome

SECONDARY OUTCOMES:
Asthma control change comparing groups | Baseline to week 16
  % of individuals with greater than or equal to 0.5 point change in ACQ6 in intervention group compared to control group. Change in score of ACQ6 (Asthma Control Questionnaire 6) in intervention group versus usual care group. Score range 0 - 36 with higher scores representing a worse outcome
Asthma Quality of Life overall change | Baseline to week 16
  Change in AQLQ score in intervention group versus usual care group. Score range 32 - 224 with lower scores representing a worse outcome
Asthma Quality of Life improvement: % | Baseline to seek 16
  % of individuals with greater than or equal to 0.5 point change in ACQ6 in intervention group compared to control group. Score range 32 - 224 with lower scores representing a worse outcome
Asthma control long term | Baseline to 52 weeks
  Change in ACQ6 score from baseline to 1 year in intervention group- Score range 0 - 36 with higher scores representing a worse outcome
Asthma quality of life long term: AQLQ score | Baseline to 52 weeks
  Change in AQLQ score
Treatment burden | Baseline to 16 weeks
  Change in asthma medication use
Treatment burden long term | Baseline to 52 weeks
  Change in asthma medication use
Healthcare use | Baseline to 16 weeks
  Change in number of unscheduled medical attendances
Healthcare use long term | Baseline to 52 weeks
  Change in number of unscheduled medical attendances

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Cowan, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

REFERENCES:
- [Derived] Sharma V, Ricketts HC, McCombie L, Brosnahan N, Crawford L, Slaughter L, Goodfellow A, Steffensen F, Buchan DS, Chaudhuri R, Lean MEJ, Cowan DC. A Total Diet Replacement Weight Management Program for Difficult-to-Treat Asthma Associated With Obesity: A Randomized Controlled Feasibility Trial. Chest. 2023 May;163(5):1026-1037. doi: 10.1016/j.chest.2023.01.015. Epub 2023 Jan 14. PMID 36649753